CLINICAL TRIAL: NCT00772278
Title: A Randomized Evaluation of Short Term and Long Term Outcome After Endovascular Repair by Stenting of Carotid Artery Stenosis in Patients With Severe (70% and Higher) Asymptomatic Carotid Stenosis
Brief Title: Comparing Carotid Stenting With Endarterectomy in Severe Asymptomatic Carotid Stenosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Dallit Manheim, Principal Investigator, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMC-07-0094-CTIL; cas vs cea-001-carmel (Other: Carmel Medical Center)
Record Dates: First submitted 2008-09-29; First posted 2008-10-15 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Carotid Stenosis
Keywords: carotid stenosis; asymptomatic; carotid stenting; carotid endarterectomy
MeSH Terms: conditions — Carotid Stenosis | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CAS (Active Comparator): carotid artery stenting
  Interventions: Procedure: carotid artery stenting
- CEA (Active Comparator): carotid endarterectomy
  Interventions: Procedure: carotid endarterectomy

INTERVENTIONS:
Procedure: carotid artery stenting — carotid artery angiography, angioplasty and stenting
  Other Names: carotid stent - precise - rapid exchange® (Cordis, FL, USA); carotid artery filter - angioguard® (Cordis, FL, USA)
  Arms: CAS
Procedure: carotid endarterectomy — open surgery including endarterectomy
  Arms: CEA

SUMMARY:
Purpose of this study:

Primary:

• Comparison of cardiovascular mortality and morbidity which includes cardiac and neurological morbidity (TIA and CVA) in the two invasive treatments of asymptomatic carotid artery stenosis

Secondary:

* Comparison of non cardiovascular morbidity caused by the two invasive techniques

  1. morbidity at the site of incision (infection or local hematoma)
  2. damage to cranial nerves (hypoglossus, vagus)
  3. brain hyperperfusion which is defined as severe headache which is not responsive to analgesics with or without nausea and vomiting.
  4. events of bradycardia within the first 24 hours, clinically evident and/or silent
* microembolic brain events immediately after the procedure and their relationship with morbidity and/or mortality due to TIA's or CVA's
* the change in the stenotic carotid artery at the time of follow up with duplex of neck arteries
* the comparison of the affect of the two procedures on patient life style

DETAILED DESCRIPTION:
Background: the surgical treatment of severe carotid artery stenosis (>70%) has been proven effective in prevention of cerebral vascular events in asymptomatic patients as compared with non invasive treatment (1, 5, 7). The currently accepted surgical treatment is called endarterectomy and includes surgery under regional and general anesthesia, in which the neck is opened, the common carotid artery, the bifurcation and the internal and external carotid artery are exposed, 5000 units of intravenous (IV) heparin is given and the arteries are occluded. The diseased artery is opened and the atherosclerotic plaque is excised, after the artery is cleaned the opening is sutured and the blood supply is reestablished. At the end of the procedure the incision is closed. The patient is transferred to recovery for four hours of surveillance, and 500 units/hour of heparin IV is started, which is continued for 12 hours. After an additional day of surveillance in the department the patient is discharged home. Two weeks after the operation the patient is invited to the out patient clinic for wound surveillance and to take out the skin staples. After which the patient is under surveillance after 3 months, 6 months, and then yearly, which involves a physical examination by a physician and a duplex examination of carotid arteries. A regiment of 100mg of Aspirin per day is initiated at the time of diagnosis. Complications associated with this procedure: a 1-3% of patients develop a transient ischemic accident (TIA) or cerebrovascular accident (CVA), cardiac complications depending on individual risk factors (0.5%), bleeding and infection at incision site is at the rate of 5%, 2-8% of patients suffer from cranial nerve damage (including hypoglossus and vagus), 2-3% of patients suffer from brain hyperperfusion, finally, stenosis recurs in 10-15% of patients.

Recently endovascular technique involving stent placement has been introduced to treat carotid artery stenosis. Early studies found this technique to be equal to traditional carotid endarterectomy in mortality and morbidity (8). Complications associated with endovascular stenting: 1-3% of patients develop a TIA or a CVA, bleeding at artery access site is at the rate of 1%, cardiac complications depending on individual risk factors (0.5%), 1-4% of patients suffer from a periprocedural arterial thromboembolic events, finally, 1% of patients suffer from renal function deterioration. Invasive treatment of carotid artery stenosis, traditional or endovascular, may be accompanied by microembolic events, which, do not necessarily result in cerebral ischemia with evident neurological deficiency. These events, however, may be noted on brain CT and may result in cognitive decline (2-4%). The role of stent deposition in conjunction with a vascular protective device, in protecting from microembolic events is still unclear.

In this study, price-rapid exchange® (Cordis, FL, USA) will be evaluated in the treatment of asymptomatic carotid artery stenosis. Traditional indications for stent placement will be used: stenosis of 70% or more demonstrated by carotid artery duplex, CTA or MRA. The stent is placed into the area of stenosed carotid artery using percutaneous approach in the operating room. The artery is visualized by injecting contrast material, a vascular protective device, angioguard® (Cordis, FL, USA), is placed downstream from carotid artery stenosis, the stent is inserted and expanded by a balloon, amiia® (Cordis, FL, USA). Furthermore, a completion angiography is preformed to visualize the final stent location and the protective vascular device is removed. A regiment of 100mg Aspirin, once daily, is initiated before endovascular treatment, and then continued as a part of a permanent treatment. Five thousand units of intravenous heparin are given at the beginning of the endovascular procedure. Heparin is than continued at 500 units per hour for the next 12 hours. The patient is discharged one day after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Stenosis of 70% or more by carotid artery duplex, CTA or MRA.
* No evidence of TIA or CVA originating in area of the brain supplied by the carotid artery under study, in the four months preceding treatment.
* Eligibility for both treatment options:

  1. suited for operative treatment as assessed by an anesthesiologist
  2. suited for endovascular procedure by established radiological guidelines (including: access to the stenotic area via the vessels of the aortic arch, the absence of occlusion preventing this access, absence of significant atherosclerosis within the arch of aorta, absence of torturous anatomy of the common and internal carotid artery, and absence of thrombus in the area of stenosis)

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2009-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
comparison of cardiovascular mortality and morbidity which includes cardiac and neurological morbidity (TIA and CVA) in the two invasive treatments of asymptomatic carotid artery stenosis | 2 years

SECONDARY OUTCOMES:
incision site morbidity | 2 years
cranial nerves damage | 2 years
brain hyperperfusion | 2 years
bradycardia within the first 24 hours | 2 years
microembolic brain events | 2 years
long term recurrence | 2 years
effect on patient life style | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dallit Mannheim, Dr., Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel